CLINICAL TRIAL: NCT03403140
Title: Multicenter Extension Study To 104 Weeks To Asses The Efficacy, Safety And Immunogenicity Of Enerceptan® In Combination With Methotrexate For The Treatment Of Patients With Rheumatoid Arthritis
Brief Title: Long Term Efficacy, Safety and Immunogenicity of Enerceptan in Rheumatoid Arthritis ( GEMENE002 )
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gema Biotech S.A. (Industry)
Collaborators: QUID Quality in Drugs and Devices Latin American Consulting SRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMENE002
Record Dates: First submitted 2017-11-30; First posted 2018-01-18 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Enerceptan®. Injectable Solution in prefilled syringes
  Source: GEMABIOTECH S. A. Formulation per unit:
  1,0 ml of Enerceptan® contains 50 mg solution of Etanercept /Once a week Methotrexate 15 to 25 mg / Once a week
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Enerceptan®. Injectable Solution in prefilled syringes
  Source: GEMABIOTECH S. A. Formulation per unit:
  1,0 ml of Enerceptan® contains 50 mg solution of Etanercept /Once a week Methotrexate 15 to 25 mg / Once a week

SUMMARY:
The purpose of this study is to asses the long term efficacy, safety and immunogenicity of ENERCEPTAN® in combination with Methotrexate for the treatment of patients with rheumatoid arthritis up to 104 weeks

DETAILED DESCRIPTION:
This is a prospective study, single treatment arm of 72 weeks of duration. Patients who completed the original study GEMENE001 may enroll in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Having completed the final active treatment visit of the GEMENE001 study, the same day or within 28 days prior to entry in this study.
2. Women of childbearing age must commit to be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of Enerceptan®. Suitable methods of contraception are oral contraceptives, IUDs, bilateral tubal ligation, vasectomy or double barrier methods such as condoms or spermicidal diaphragm, sponge, contraceptive foam or gel, heterosexual abstinence. Men should not conceive up to 12 weeks after stopping the MTX
3. Informed consent must be signed before making any study-specific procedure

Exclusion Criteria:

1. Have temporarily interrupted the investigational product in the final study visit GEMENE001 and, according to the investigator's opinion, this represents an unacceptable risk to the patient whether this participates in the GEMENE002 study.
2. Simultaneous treatment with other investigational drug or participation in another clinical study that the investigator considers inadvisable.
3. Women who are pregnant or breastfeeding.
4. History of lack of response or loss of response to previous therapy with Etanercept in the GEMENE001 study.
5. Chronic antibiotic therapy, if the investigator considers this may affect the safety of the subject or the assessment of the study results.
6. Any previous or current serious medical conditions which had appeared during the study GEMENE001 that, in the opinion of the investigator, constitute a contraindication for the study treatment, as:
7. Administration of vaccines:

   1. Subjects who have received a live attenuated vaccine within 3 months prior to the selection Visit (for example, varicella-zoster, oral polio, rabies, yellow fever vaccines.)
   2. Subjects who have received the BCG vaccine within the GEMENE001 study
8. Presence of :

   a. At the time of the inclusion i. Active infections. ii. Fever (≥38 °C) or active, chronic or recurrent infections that require treatment with antibiotics, antiviral, or anti-fungal drugs within 4 weeks prior to Screening Visit, or history of frequent recurrent infections unacceptable to the investigator's opinion.

   iii. Non-healing infected skin ulcers. b. In the previous time: i. Background of recurrent bacterial, viral, fungal (excluding superficial infections or nail bed mycosis), mycobacterial or other severe infections within the last month previous to selection.

   ii. Hospitalization for infection or Subjects who have received antibiotics intravenously within the last month or orally within the last 2 weeks.

   iii. Subjects with herpes zoster in the last 2 months.
9. Past history of drug or alcohol abuse within the study GEMENE001.
10. Any condition that, in the investigator's opinion, would not allow compliance with the guidelines of the study by the patient.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 72 weeks
  Infections, hematological disorders,.neurologic disorders and malignancies .

SECONDARY OUTCOMES:
Lab tests alterations [Safety and Tolerability]). | 72 weeks
  Serum Hematological and chemistry values
Local reactions [Safety and Tolerability]). | 72 weeks
  Incidence, description and severity of Local Adverse Drug Reactions
ACR20 | 20 and 72 Weeks
  ACR (American College of Rheumatology) 20 The percentage of patients who achieved ACR20 at Week 32 is the primary end point. Signs and symptoms are assessed with a composite rating scale of the ACR (American College of
  Rheumatology) that includes 7 variables:
  * Tender Joints Count
  * Swollen Joints Count
  * Levels of an acute phase reactant (CRP level)
  * Patient's assessment of pain
  * Patient's global assessment of disease activity
  * Physician's global assessment of disease activity
  * Patient's assessment of physical function
ACR50 | 20 and 72 Weeks
  ACR50 is defined as the percentage of patients who achieve at least 50% improvement in both tender joint count and swollen joint count, and at least 50% improvement in at least 3 of the 5 other assessments.
ACR70 | 20 and 72 Weeks
  ACR70 is defined as the percentage of patients who achieve at least 70% improvement in both tender joint count and swollen joint count, and at least 50% improvement in at least 3 of the 5 other assessments.
DAS (Disease activity state) | 20 and 72 Weeks
  It will be measured using the DAS (Disease activity state) 28. DAS28 is a composite score that includes 4 variables:
  * Tender Joints Count (based on 28 joints)
  * Swollen Joints Count (based on 28 joints)
  * Patient's global assessment of disease activity
  * Marker of inflammation: C REACTIVE PROTEIN
Change in modified van der Heijde Sharp score | 20 and 72 Weeks
  The Sharp method is a composite X-ray scoring system used to assess structural (joint) disease progression in rheumatoid arthritis. The method evaluates both joint erosions (JE) and joint space narrowing (JSN) in bilateral hand and foot joints. The Sharp/van der Heijde method assesses erosions and joint space narrowing separately in the hands and feet, and has a range from 0 to 448. Thirty-two joints in the hands and 12 in the feet are scored for erosions, with a maximum score of five per joint in the hands and 10 per joint in the feet. Joint space narrowing is graded from 0 to 4 in 30 joints in the hands and in 12 joints in the feet.
  The principal score used in the analyses is the total score, which is the sum of the erosion score and the joint space narrowing score.
Physical function | 20 and 72 Weeks
  Improvement in physical function is assessed by change from baseline in HAQ (Health Assessment Questionnaire).The HAQ-DI (disability index) is composed of 8 categories as follows: dressing and grooming, arising, eating, walking, hygiene, reach, grip and activities, for which there are at least 2 questions by category. The patient will be asked to score how difficult he/she feels it is to perform such activities using a 0 to 3 scoring (0=without any difficulty,
  1=with some difficulty, 2=with much difficulty and 3=unable to do). If the patient is using assistance for any of these activities, scoring may be adjusted. For each category, the highest score given for one of the question is attributed to the category. The total score is the sum of all categories' scores divided by the number of answered categories (at least 3 categories should be answered)
Functional Assessment of Chronic Illness Therapy Fatigue scale (FACIT-Fatigue) | 20 and 72 Weeks
  The FACIT-Fatigue is a 13-item questionnaire rated 0 to 4. The patient will be asked to answer to 13 questions rated 0 to 4 (0=not at all,
  1=a little bit, 2=some what, 3=quite a bit, 4=very much
Steady state concentration | 20 and 72 Weeks
  Etanercept concentration measure
Immunogenicity | 20 and 72 Weeks
  Antibodies anti-Etanercept measure

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Medico CER, Bs As, Argentina

IPD SHARING:
Plan to Share IPD: Undecided